CLINICAL TRIAL: NCT03443843
Title: A Double-Blind Placebo-Controlled Crossover Study to Evaluate Objective Changes in Nasal Airflow of Loratadine/Pseudoephedrine Tablet and Fluticasone Propionate Nasal Spray in Subjects Following Allergen Exposure in an Environmental Exposure Unit
Brief Title: A Study to Evaluate Changes in Nasal Airflow of Loratadine/Pseudoephedrine Tablet and Fluticasone Propionate Nasal Spray in Subjects Following Allergen Exposure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19880
Record Dates: First submitted 2018-02-20; First posted 2018-02-23 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Loratadine; Acetaminophen; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Treatment phase will consist of four treatment visits separated by 14 (+/- 1) days between visits. Each treatment sequence consists of a single dose of each of the 4 treatments.
  Interventions: Drug: loratadine + pseudoephedrine sulfate (BAY818725/Claritin-D); Drug: Placebo tablet; Drug: Fluticasone Propionate; Drug: Placebo spray
- Sequence 2 (Experimental): Treatment phase will consist of four treatment visits separated by 14 (+/- 1) days between visits. Each treatment sequence consists of a single dose of each of the 4 treatments.
  Interventions: Drug: loratadine + pseudoephedrine sulfate (BAY818725/Claritin-D); Drug: Placebo tablet; Drug: Fluticasone Propionate; Drug: Placebo spray
- Sequence 3 (Experimental): Treatment phase will consist of four treatment visits separated by 14 (+/- 1) days between visits. Each treatment sequence consists of a single dose of treatment each of the 4 treatments.
  Interventions: Drug: loratadine + pseudoephedrine sulfate (BAY818725/Claritin-D); Drug: Placebo tablet; Drug: Fluticasone Propionate; Drug: Placebo spray
- Sequence 4 (Experimental): Treatment phase will consist of four treatment visits separated by 14 (+/- 1) days between visits. Each treatment sequence consists of a single dose of treatment each of the 4 treatments.
  Interventions: Drug: loratadine + pseudoephedrine sulfate (BAY818725/Claritin-D); Drug: Placebo tablet; Drug: Fluticasone Propionate; Drug: Placebo spray

INTERVENTIONS:
Drug: loratadine + pseudoephedrine sulfate (BAY818725/Claritin-D) — Single dose of Loratadine/pseudoephedrine in tablet 5 mg/120 mg orally
Drug: Placebo tablet — Placebo tablet orally
Drug: Fluticasone Propionate — Fluticasone Propionate Nasal Spray 50mcg per spray, 2 sprays per nostril
Drug: Placebo spray — Placebo Nasal Spray, 2 sprays per nostril

SUMMARY:
The purpose of the study is to evaluate changes in nasal airflow caused by loratadine 5 mg/pseudoephedrine sulfate 120 mg (Claritin D) tablet and fluticasone propionate 50 mcg per spray nasal spray (Flonase) in subjects suffering from nasal congestion and other allergy symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory male and female subjects between 18 to 65 years of age
* Self-reported seasonal allergic rhinitis to ragweed pollen for at least 2 years prior to screening
* Documented positive skin prick test response to common ragweed (ambrosia artemisiifolia) pollen at screening or within the previous 12 months conducted at research site (prick with wheal diameter >= 5 mm larger than the diluent response)
* In order to qualify to continue to treatment phase, at the end of priming phase (which is 3 hours), Total Symptom Score (TSS) has to be ≥ 7, with nasal congestion score alone ≥ 2 and change in peak nasal inspiratory flow (PNIF) has to be ≥ 15% from pre-prime baseline;
* Subject is willing to stop use of current decongestant and allergy medications at the start of the washout period prior to priming and during the trial
* At the discretion of the investigators, subjects may be considered with self-reported mild intermittent asthma (Using <=2 doses of SABA (short-acting beta agonists) per week) or exercise-induced asthma
* Subject is free of any clinically significant disease that required a physician´s care and/or would interfere with trial evaluations, procedures or participation
* Subject is able to repeatedly and reliably perform PNIF measurements and must achieve PNIF value of >=60L/min at screening
* Subject must be capable of reading English and willing to participate in all aspects of the study

Exclusion Criteria:

- Any significant medical condition which, in the judgment of the investigator, is a contraindication to the use of loratadine, pseudoephedrine and fluticasone propionate, or might interfere with the trial. These may include subjects with injury or surgery to the nose that is not fully healed, fungal infections, immunocompromised conditions (HIV, tuberculosis), severe nosebleeds, narrow-angle glaucoma, chickenpox measles..., severe facial pain or thick nasal discharge, sinusitis, constant whistling sound from the nose, structured abnormality of the nose, uncontrolled thyroid disease (e.g., hyperthyroidism, hypothyroidism), uncontrolled diabetes mellitus, coronary heart disease ischemic heart disease, uncontrolled high blood pressure, symptomatic prostatic hypertrophy, bladder neck obstruction, hepatic insufficiency, renal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Average percent change in PNIF (Peak Nasal Inspiratory Flow) from 0 to 4 hours after dosing | Up to 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Ng CC, Romaikin D, Steacy LM, Stevens DA, Walker TJ, Adams DE, Ellis AK. Comparative nasal airflow with loratadine-pseudoephedrine and fluticasone nasal spray for allergic rhinitis. Ann Allergy Asthma Immunol. 2021 Sep;127(3):342-348.e2. doi: 10.1016/j.anai.2021.05.001. Epub 2021 May 14. PMID 34000435